CLINICAL TRIAL: NCT02200887
Title: Role of Sleep Homeostasis in the Development of the L-Dopa Induced Dyskinesias in Patients With Parkinson's Disease
Brief Title: Sleep Homeostasis in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Salvatore Galati (Other Government)
Responsible Party: Sponsor-Investigator, Salvatore Galati, MD, head of service, Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Other Study IDs: EOC-NSI.12.01
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
Keywords: Dyskinesia; Slow Wave Sleep
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Advanced Parkinsons Disease: Polysomnogram
- Parkinsons Disease with Dyskinesia: Polysomnogram
- De novo Parkinsons Disease: Polysomnogram
- Healthy Volunteers: Polysomnogram

SUMMARY:
Parkinson's disease is characterized in the advanced phases by an altered response to dopaminergic therapy for the occurrence of abnormal movements called dyskinesias, that worsens the quality of life of the patient and exposes him to comorbidities. Several data show a reduction in the amount of slow wave sleep that correlates inversely with disease duration. Since this stage of sleep is linked to mechanisms of deletion of superfluous information the investigators hypothesize that the onset of dyskinesias is related to such alteration of sleep.

-This study is aimed to investigate, by means of high-density electroencephalography (hd-EEG), the sleep and in particular the slow wave in order to clarify the relations with the development of dyskinesias.

DETAILED DESCRIPTION:
Wakefulness in PD is frequently interrupted by sleep episodes, even rapid eye movement sleep (REM), whilst nocturnal sleep is disturbed by abnormal motor activity interference, such as REM sleep behaviour disorder (RBD) or periodic limb movements (PLMS). Several lines of evidence have suggested a close relation between sleep-wake changes and dopaminergic degeneration in PD(1-7) while sleep disorders commonly precede the clinical motor onset by many years (8,9). On the other hand, morning motor performance improvement is frequently mentioned by patients, mainly in those with long disease duration and motor fluctuation (10,11). Of note, the same state of vigilance can profoundly influence some clinical PD features (for instance rigidity) as well as basal ganglia neuronal activity(12).

Few reports have shown changes in sleep architecture: a reduction of the amount of SWS in parallel with disease duration (13-15) has been observed, but no study, so far, has addressed how sleep may impact on LID. Once these abnormal movements develop, they are difficult to treat and negatively affect the quality of life and the treatment costs of PD patients (16,17). Although levodopa represents, so far, the more effective treatment for PD patients (18,19) to ameliorate the cardinal signs such as bradykinesia/akinesia and rigidity (20), as the disease progresses, these benefits are in some measure abolished by the emergence of dyskinesia (21). During the early stages PD patients experience a rather satisfying quality of life that is impeded in the advanced stages by the emerging of these involuntary movements frequently at the peak of the levodopa effect (16,22,23). In other words, when the patients experience these motor complications (shortening motor response and development of dyskinesia) the delivery of levodopa without inducing dyskinesia becomes increasingly difficult (21,24-27).

Several efforts have been made in order to find "pure" anti-dyskinetic drugs that are able to uncouple the anti-akinetic effect from the dyskinetic response. Serotoninergic receptor agonists were claimed to be drugs against dyskinesia (28), however, it was observed that they may also impair levodopa efficacy (29-31). As of today, no clinical effective therapies are able to alleviate dyskinesia without worsening parkinsonism.

Great efforts have been made to clarify LID pathogenesis, emphasizing the role of pulsative stimulation of striatal receptors by dopaminergic treatment (25) and more recently, on molecular changes of postsynaptic (32,33) or presynaptic mechanisms (34). Although no conclusive results on LID pathogenesis have been achieved, indeed disease duration (i.e. the degree of dopaminergic degeneration) rather than long-term use of levodopa, seems to play a crucial role (22,23). This notion can be inferred from clinical practice, but is also evident in MPTP-induced parkinsonism in humans in which the extended dopaminergic lesion caused within a few days the development of dyskinesias undistinguishable from those in the idiopathic form (35).

General Aim:

The study is aimed 1) to define abnormal cortical synaptic homeostasis, measured by means of SWS and waking EEG evoked responses, as key components for the development of LID; 2) to analyse the impact of anti-dyskinetic effect of rTMS on the SWA in additional ten PD patient with LID.

Specific aims:

1. To compare, in the four groups of subjects (control, de novo, advanced without dyskinesia, and advanced with dyskinesia), changes of the EEG features of NREM sleep: slow wave/slow oscillation and sleep spindles. A significant reduction of the physiological reduction of SWA in dyskinetic patients in comparison with the other groups is expected.
2. To identify the homeostatic reduction of cortical synaptic strength (downscaling) in the four categories of subjects by comparing late sleep (i.e. towards morning) SWA with early sleep (i.e. at the beginning of the night) SWA as well as by comparing the overnight changes in the amplitude of EEG somatosensory, auditory and visual evoked responses recorded before and after sleep. The study is aimed to demonstrate the reduction/absence of a physiological downscaling in dyskinetic patients versus the other groups.
3. To analyse the effect of rTMS on SWA of PD patients with LID in order to demonstrate a recovery of physiological downscaling of SWA in these patients parallel to the reduction of dyskinesia.

ELIGIBILITY:
Inclusion Criteria:

* clinical characteristics of the patients must be according the UK (United Kingdom) Brain Bank

Exclusion Criteria:

* anamnestic obstructive sleep apneas syndrome
* known cognitive deterioration or with MMSE (Mini-Mental State Examination) ≤24/30
* depression ≥ 20 of the BDI scale (Beck Depression Inventory)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with parkinson disease
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Slow wave sleep | 1 night
  Percentage of total sleep classified as slow wave sleep

SECONDARY OUTCOMES:
Amplitude of slow waves during sleep | 1 Night
  Reduction of homeostatic synaptic plasticity during the time of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Galati, MD, Principal Investigator — Ospedale Regionale di Lugano
Locations (1):
- Ospedale Regionale di Lugano, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Background] Poewe W, Hogl B. Parkinson's disease and sleep. Curr Opin Neurol. 2000 Aug;13(4):423-6. doi: 10.1097/00019052-200008000-00009. No abstract available. PMID 10970059
- [Background] Rye DB, Jankovic J. Emerging views of dopamine in modulating sleep/wake state from an unlikely source: PD. Neurology. 2002 Feb 12;58(3):341-6. doi: 10.1212/wnl.58.3.341. No abstract available. PMID 11839829
- [Background] Moller JC, Rethfeldt M, Korner Y, Stiasny-Kolster K, Cassel W, Meindorfner C, Rissling I, Kruger HP, Oertel WH. Daytime sleep latency in medication-matched Parkinsonian patients with and without sudden onset of sleep. Mov Disord. 2005 Dec;20(12):1620-2. doi: 10.1002/mds.20630. PMID 16078226
- [Background] Moller JC, Unger M, Stiasny-Kolster K, Kaussner Y, Penzel T, Oertel WH, Hemmeter U. Continuous sleep EEG monitoring in PD patients with and without sleep attacks. Parkinsonism Relat Disord. 2009 Mar;15(3):238-41. doi: 10.1016/j.parkreldis.2008.05.009. Epub 2008 Jul 10. PMID 18619893
- [Background] Valko PO, Waldvogel D, Weller M, Bassetti CL, Held U, Baumann CR. Fatigue and excessive daytime sleepiness in idiopathic Parkinson's disease differently correlate with motor symptoms, depression and dopaminergic treatment. Eur J Neurol. 2010 Dec;17(12):1428-36. doi: 10.1111/j.1468-1331.2010.03063.x. PMID 20491889
- [Background] Benninger DH, Michel J, Waldvogel D, Candia V, Poryazova R, van Hedel HJ, Bassetti CL. REM sleep behavior disorder is not linked to postural instability and gait dysfunction in Parkinson. Mov Disord. 2010 Aug 15;25(11):1597-604. doi: 10.1002/mds.23121. PMID 20629146
- [Background] Unger MM, Belke M, Menzler K, Heverhagen JT, Keil B, Stiasny-Kolster K, Rosenow F, Diederich NJ, Mayer G, Moller JC, Oertel WH, Knake S. Diffusion tensor imaging in idiopathic REM sleep behavior disorder reveals microstructural changes in the brainstem, substantia nigra, olfactory region, and other brain regions. Sleep. 2010 Jun;33(6):767-73. doi: 10.1093/sleep/33.6.767. PMID 20550017
- [Background] Claassen DO, Josephs KA, Ahlskog JE, Silber MH, Tippmann-Peikert M, Boeve BF. REM sleep behavior disorder preceding other aspects of synucleinopathies by up to half a century. Neurology. 2010 Aug 10;75(6):494-9. doi: 10.1212/WNL.0b013e3181ec7fac. Epub 2010 Jul 28. PMID 20668263
- [Background] Bassetti CL. Nonmotor disturbances in Parkinson's disease. Neurodegener Dis. 2011;8(3):95-108. doi: 10.1159/000316613. Epub 2010 Dec 23. PMID 21196687
- [Background] Currie LJ, Bennett JP Jr, Harrison MB, Trugman JM, Wooten GF. Clinical correlates of sleep benefit in Parkinson's disease. Neurology. 1997 Apr;48(4):1115-7. doi: 10.1212/wnl.48.4.1115. PMID 9109914
- [Background] Bateman DE, Levett K, Marsden CD. Sleep benefit in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1999 Sep;67(3):384-5. doi: 10.1136/jnnp.67.3.384. No abstract available. PMID 10449564
- [Background] Stefani A, Galati S, Peppe A, Bassi A, Pierantozzi M, Hainsworth AH, Bernardi G, Orlacchio A, Stanzione P, Mazzone P. Spontaneous sleep modulates the firing pattern of parkinsonian subthalamic nucleus. Exp Brain Res. 2006 Jan;168(1-2):277-80. doi: 10.1007/s00221-005-0175-y. Epub 2005 Nov 18. PMID 16328297
- [Background] Diederich NJ, Vaillant M, Mancuso G, Lyen P, Tiete J. Progressive sleep 'destructuring' in Parkinson's disease. A polysomnographic study in 46 patients. Sleep Med. 2005 Jul;6(4):313-8. doi: 10.1016/j.sleep.2005.03.011. PMID 15946897
- [Background] Romigi A, Placidi F, Peppe A, Pierantozzi M, Izzi F, Brusa L, Galati S, Moschella V, Marciani MG, Mazzone P, Stanzione P, Stefani A. Pedunculopontine nucleus stimulation influences REM sleep in Parkinson's disease. Eur J Neurol. 2008 Jul;15(7):e64-5. doi: 10.1111/j.1468-1331.2008.02167.x. Epub 2008 May 15. No abstract available. PMID 18484989
- [Background] Dodel RC, Berger K, Oertel WH. Health-related quality of life and healthcare utilisation in patients with Parkinson's disease: impact of motor fluctuations and dyskinesias. Pharmacoeconomics. 2001;19(10):1013-38. doi: 10.2165/00019053-200119100-00004. PMID 11735671
- [Background] Devos D; French DUODOPA Study Group. Patient profile, indications, efficacy and safety of duodenal levodopa infusion in advanced Parkinson's disease. Mov Disord. 2009 May 15;24(7):993-1000. doi: 10.1002/mds.22450. PMID 19253412
- [Background] Mercuri NB, Bernardi G. The 'magic' of L-dopa: why is it the gold standard Parkinson's disease therapy? Trends Pharmacol Sci. 2005 Jul;26(7):341-4. doi: 10.1016/j.tips.2005.05.002. PMID 15936832
- [Background] Poewe W, Antonini A, Zijlmans JC, Burkhard PR, Vingerhoets F. Levodopa in the treatment of Parkinson's disease: an old drug still going strong. Clin Interv Aging. 2010 Sep 7;5:229-38. doi: 10.2147/cia.s6456. PMID 20852670
- [Background] Katzenschlager R, Lees AJ. Treatment of Parkinson's disease: levodopa as the first choice. J Neurol. 2002 Sep;249 Suppl 2:II19-24. doi: 10.1007/s00415-002-1204-4. PMID 12375059
- [Background] Jankovic J, Stacy M. Medical management of levodopa-associated motor complications in patients with Parkinson's disease. CNS Drugs. 2007;21(8):677-92. doi: 10.2165/00023210-200721080-00005. PMID 17630819
- [Background] Nadjar A, Gerfen CR, Bezard E. Priming for l-dopa-induced dyskinesia in Parkinson's disease: a feature inherent to the treatment or the disease? Prog Neurobiol. 2009 Jan 12;87(1):1-9. doi: 10.1016/j.pneurobio.2008.09.013. Epub 2008 Sep 30. PMID 18938208
- [Background] Berthet A, Bezard E. Dopamine receptors and L-dopa-induced dyskinesia. Parkinsonism Relat Disord. 2009 Dec;15 Suppl 4:S8-12. doi: 10.1016/S1353-8020(09)70827-2. PMID 20123563
- [Background] Melamed E, Zoldan J, Galili-Mosberg R, Ziv I, Djaldetti R. Current management of motor fluctuations in patients with advanced Parkinson's disease treated chronically with levodopa. J Neural Transm Suppl. 1999;56:173-83. doi: 10.1007/978-3-7091-6360-3_11. PMID 10370911
- [Background] Olanow CW, Obeso JA, Stocchi F. Continuous dopamine-receptor treatment of Parkinson's disease: scientific rationale and clinical implications. Lancet Neurol. 2006 Aug;5(8):677-87. doi: 10.1016/S1474-4422(06)70521-X. PMID 16857573
- [Background] Antonini A, Ursino G, Calandrella D, Bernardi L, Plebani M. Continuous dopaminergic delivery in Parkinson's disease. J Neurol. 2010 Nov;257(Suppl 2):S305-8. doi: 10.1007/s00415-010-5714-1. PMID 21080194
- [Background] Stefani A, Galati S, Brusa L, Pierantozzi M, Peppe A, Stanzione P. Pathological gambling from dopamine agonist and deep brain stimulation of the nucleus tegmenti pedunculopontine. BMJ Case Rep. 2010 Nov 18;2010:bcr0220102774. doi: 10.1136/bcr.02.2010.2774. PMID 22798481
- [Background] Munoz A, Li Q, Gardoni F, Marcello E, Qin C, Carlsson T, Kirik D, Di Luca M, Bjorklund A, Bezard E, Carta M. Combined 5-HT1A and 5-HT1B receptor agonists for the treatment of L-DOPA-induced dyskinesia. Brain. 2008 Dec;131(Pt 12):3380-94. doi: 10.1093/brain/awn235. Epub 2008 Oct 24. PMID 18952677
- [Background] Olanow CW, Kieburtz K, Stern M, Watts R, Langston JW, Guarnieri M, Hubble J; US01 Study Team. Double-blind, placebo-controlled study of entacapone in levodopa-treated patients with stable Parkinson disease. Arch Neurol. 2004 Oct;61(10):1563-8. doi: 10.1001/archneur.61.10.1563. PMID 15477510
- [Background] Huot P, Fox SH, Brotchie JM. The serotonergic system in Parkinson's disease. Prog Neurobiol. 2011 Oct;95(2):163-212. doi: 10.1016/j.pneurobio.2011.08.004. Epub 2011 Aug 22. PMID 21878363
- [Background] Jenner P. Functional models of Parkinson's disease: a valuable tool in the development of novel therapies. Ann Neurol. 2008 Dec;64 Suppl 2:S16-29. doi: 10.1002/ana.21489. PMID 19127585
- [Background] Calabresi P, Di Filippo M, Ghiglieri V, Tambasco N, Picconi B. Levodopa-induced dyskinesias in patients with Parkinson's disease: filling the bench-to-bedside gap. Lancet Neurol. 2010 Nov;9(11):1106-17. doi: 10.1016/S1474-4422(10)70218-0. Epub 2010 Sep 27. PMID 20880751
- [Background] Galati S, Stanzione P, D'Angelo V, Fedele E, Marzetti F, Sancesario G, Procopio T, Stefani A. The pharmacological blockade of medial forebrain bundle induces an acute pathological synchronization of the cortico-subthalamic nucleus-globus pallidus pathway. J Physiol. 2009 Sep 15;587(Pt 18):4405-23. doi: 10.1113/jphysiol.2009.172759. Epub 2009 Jul 21. PMID 19622605
- [Background] Langston JW, Ballard P. Parkinsonism induced by 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine (MPTP): implications for treatment and the pathogenesis of Parkinson's disease. Can J Neurol Sci. 1984 Feb;11(1 Suppl):160-5. doi: 10.1017/s0317167100046333. PMID 6608979